CLINICAL TRIAL: NCT05550077
Title: Optical Coherence Tomography for Intracranial Atherosclerotic Stenosis: a Prospective Registry Study (OCT-ICAS)
Brief Title: Optical Coherence Tomography for Intracranial Atherosclerotic Stenosis
Acronym: OCT-ICAS
Status: Recruiting | Type: Observational
Sponsor: jiaoliqun (Other)
Responsible Party: Sponsor-Investigator, jiaoliqun, Director, Department of Interventional Neuroradiology, Principal Investigator, Clinical Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Other Study IDs: OCT-ICAS
Record Dates: First submitted 2022-09-18; First posted 2022-09-22 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Intracranial Atherosclerosis; Optical Coherence Tomography; Plaque, Atherosclerotic; Artery Stenosis; Ischemic Stroke
Keywords: Optical Coherence Tomography; Intravascular Imaging; Intracranial Atherosclerotic Stenosis; Percutaneous Transluminal Angioplasty and Stenting
MeSH Terms: conditions — Intracranial Arteriosclerosis; Plaque, Atherosclerotic; Ischemic Stroke | interventions — Tomography, Optical Coherence; Angioplasty; Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Optical Coherence Tomography (OCT): OCT and other classical imaging evaluation such as Transcranial Color Doppler (TCCD) and High resolution-MRI will be performed. The tailored treatment (such as anti-thrombotic management, post-dilation, et al) will be considered when specific plaque characteristics (including but not limited to in situ thrombus formation, macrocacilfication, et al), were observed under OCT.
  Interventions: Diagnostic Test: Optical Coherence Tomography; Procedure: Percutaneous transluminal angioplasty and stenting
- Non-Optical Coherence Tomography (N-OCT): Classical imaging evaluation such as TCCD and High resolution-MRI will be performed, followed by standard percutaneous transluminal angioplasty and stenting.
  Interventions: Procedure: Percutaneous transluminal angioplasty and stenting

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography — Intravascular evaluation for vessel wall structure of intracranial atherosclerotic stenosis by application of optical coherence tomography
  Groups: Optical Coherence Tomography (OCT)
Procedure: Percutaneous transluminal angioplasty and stenting — Percutaneous transluminal angioplasty and stenting will be performed follow the standard or adjusted according to OCT evaluation.

SUMMARY:
To evaluate the clinical significance of optical coherence tomography (OCT) in interventional treatment of intracranial atherosclerotic stenosis (ICAS).

DETAILED DESCRIPTION:
Stroke was the second leading cause of death worldwide and the leading cause of death in China in 2017. ICAS accounted for 10% to 15% of ischemic stroke in Western countries, and as much as 46.6%in Asia in 2009.

For patients with ICAS, the risk of stroke is highly related to the histopathology of atheromatous plaques. Therefore, characterizing the morphology and composition of plaques in ICAS may help to predict the risk of stroke occurrence and allow the adoption of preventive or therapeutic management to prevent such life-threatening events. OCT, with a resolution of 10μm, may provide more reliable information in characterizing atheromatous plagues.

This study aims to get a better insight into the value of OCT in evaluating the vessel wall structure and therefore guiding the interventional therapy of ICAS. In addition, the clinical and biological information will be included to achieve correlation analysis so as to get biomarkers subject to various plaque characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic ICAS. Participants with ICAS with a transient ischaemic attack (TIA) or stroke attributable to the territory of the stenotic artery were defined as symptomatic. A TIA was defined as a transient episode of neurological dysfunction (focal weakness or language disturbance, transient monocular blindness, or required assistance in walking) caused by focal brain or retinal ischaemia that lasted for at least 10 minutes but resolved within 24 hours
* Stenotic degree ≥ 50%, measured by digital subtraction angiography
* The stenosis must located in at least one major intracranial artery (internal carotid artery, vertebral artery, middle cerebral artery, or basilar artery)

Exclusion Criteria:

* Arteriovenous Malformation
* Aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (aged over 18) with symptomatic ICAS (≥ 50%) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety outcomes: short-term death or stroke | 30 days after enrollment
  We defined 'short-term' as the periprocedural period, or mean follow-up time less than or equal to three months after enrollment. Stroke was identified in the vascular territory of the stenosed vessel, either ischaemic or haemorrhagic. We defined death or stroke as a composite of death of any cause or non-fatal stroke of any type in any territory.

SECONDARY OUTCOMES:
Death or stroke | 1 year after enrollment
  (long term; more than three months)
Ipsilateral stroke | 1 year after enrollment
  (same territory as the index stenosis)
Type of recurrent event | 1 year after enrollment
  (TIA, ischaemic stroke, haemorrhagic stroke)
Death | 1 year after enrollment
  (long term; more than three months)
Restenosis | 1 year after enrollment
  (≥ 50%) of the involved vessel documented by conventional cerebral angiography
Dependency | 1 year after enrollment
  Modified Rankin Scale or equivalent

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li T, Xu R, Ma Y, Wang T, Yang B, Jiao L. Calcification is a risk factor for intracranial in-stent restenosis: an optical coherence tomography study. J Neurointerv Surg. 2024 Aug 14;16(9):897-901. doi: 10.1136/jnis-2023-020624. PMID 37536931